# Informed Consent Form Cover Page for ClinicalTrials.Gov Record

## **Official Study Title:**

Sub-study: Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Brief Title:** 

A+ Treatment/Feasibility of Adapted ESDM-informed Caregiver Coaching Delivered Remotely for Children With ASD and ADHD

#### NCT #: NCT05417607

Duke University Health System (DUHS) Protocol #: Pro00085179

Document Version Date (DUHS IRB Reference Date of Consent Form): 20-SEP-2021

Document Name/Consent Type: A+ Treatment/Feasibility (Sub-study) Consent (Child participant and Adult/Parent)



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

## **Concise Summary**

The purpose of this research study is to evaluate the feasibility of an adapted Early Start Denver Model (ESDM)-informed caregiver coaching behavioral intervention. The study is being done with children who are diagnosed with both Autism Spectrum Disorder (ASD) and Attention-Deficit/Hyperactivity Disorder (ADHD), and who are between 3 and 10 years of age.

If you and your child participate, you will complete eight sessions of ESDM-informed caregiver coaching delivered weekly for 8 consecutive weeks. Sessions are done remotely and strategies are implemented within the child's typical daily routines by the caregiver.

No ADHD medication is provided by the study. The study will document whether or not your child is taking an ADHD medication prescribed by their own personal provider.

Participants will first complete screening that includes a diagnostic and behavioral assessment, collection of medical and behavioral information, questionnaires, and activities measuring attention and social interaction.

The risks of this study are minimal, which means they are not expected to be more than what is typically encountered in routine physical and psychological exams. The main risks of this study are possible fatigue or boredom from the questionnaires and assessments. Some questions asked through interviews or surveys may cause parents or children to feel uncomfortable. You can take breaks at any time and you may refuse to answer any question. There is also a risk of loss of confidentiality when participating in research.

Potential benefits: Your child may benefit by receiving diagnostic and cognitive evaluations that are conducted as part of this study. Your family could also benefit from the ESDM-based caregiver coaching.

If you are interested in learning more about this study, please continue to read below.

## INTRODUCTION

You and your child are being asked to take part in this research study because your child is part of the Duke Autism Center of Excellence ("Duke ACE Center") research program and you have expressed interest participating in the feasibility A+ Treatment study for children with ASD and ADHD.

Please read this consent form carefully and take your time making a decision. The nature of the study, including the risks and benefits, are explained below. Please ask the staff member who provided this consent form to explain any words or information that you do not clearly understand.


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

Participation in a research study is always completely voluntary. If you do agree to have your child participate, you can change your mind and may withdraw your child from the study at any time. Any services that your child receives through a Duke University-affiliated (or non-Duke affiliated) clinic or primary care provider will not be affected by your decision about your child's participation in this study. We encourage you to talk with your family and friends before you and your child decide to take part in this research study. Please tell the study doctor or study staff if your child is in another research study.

This part of the Duke ACE Center program is called the "A+ Treatment Study" and it is overseen by Dr. Lauren Franz. The A+ Treatment Project and the Duke ACE Center are sponsored by a grant from the National Institutes of Health (NIH). Portions of Dr. Franz's and the research team's salaries are paid by this grant.

#### WHO WILL BE MY CHILD'S DOCTOR ON THIS STUDY?

If you and your child decide to participate, Dr. Franz, or one of the other study doctors will be your child's study doctor.

#### WHY IS THIS STUDY BEING DONE?

Approximately half of children with ASD also have ADHD. We are studying whether it is feasible to provide an ESDM-adapted caregiver coaching intervention, remotely, with children who have both ASD and ADHD, and their caregiver(s). By studying the feasibility of this intervention, we will able to look at whether this can be done by other therapists and study teams in similar settings, and to study this particular type of intervention further.

Since many children who have ADHD also take medication for these symptoms, the study will document which children are on a stimulant medication, and which are not, so we can better understand any differences. One goal main of this research is to help doctors in the future better treat and help children with both ASD and ADHD.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Approximately 35 children and their parent(s) will take part in this study at Duke.


#### WHAT IS INVOLVED IN THE STUDY?

If you agree for you and your child to be in this study, you will be asked to sign and date this consent form electronically. The Duke A+ Treatment study will evaluate your child's health, social and language abilities, and how they interact with you and play. There will be 8 weekly coaching sessions done remotely through a teleconference platform (Zoom). Study activities will happen weekly for the first 9 weeks, and there will be a follow up time point at week 16. The visits and study activities are described below.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

Before the start of the study, our study team will complete diagnostic and cognitive assessments and interviews with you and your child to determine if your child is eligible for A+ Treatment. If your child is eligible and you and your child wish to participate, then your child will be enrolled into the study.

**Baseline Visit**: Before your first coaching session, the study team will do a brief call (10-30 minutes) with you to explain what the ESDM-informed coaching will look like and what it involves. You will also be asked to complete:

- A few surveys about your child's symptoms, health, well-being, medications, medical history, and overall functioning.
- Questionnaires about your own experiences and feelings.
- An interview and questionnaire with a study clinician or staff.
- Guided interactive tasks at home that you complete with your child, including an
  assessment of your child's behavior delivered on a smart phone or tablet, and a playbased parent-child interaction task.

**Weeks 1- 8**: Each week, you will be scheduled for a caregiver coaching session of approximately 1 hour with a study clinician. This will include setting goals together, practicing strategies, and may also include questions about how you are applying the coaching at home. You will be able to practice what you learn through coaching at home with your child during daily activities. Additionally:

 We will ask about your child's wellbeing, health, and any changes to medical history or medications.

**Week 9**: Interviews, surveys and study activities you did at the Baseline Visit will be repeated. We will also ask you questions about your experiences, feelings and opinions, related to the intervention.

## Early Start Denver Model (ESDM) - Informed Caregiver Coaching

A therapist trained in caregiver coaching of ESDM will meet with you and your child 8 times by Zoom, once a week, for about 60 minutes to coach you in the use of strategies to promote social and language abilities and behavioral regulation (e.g., reduce tantrums). Another family member may also attend these sessions, but it is important that you come to each therapy visit. This is to ensure that you learn how all the different ESDM-informed caregiver coaching strategies work together and so that you and the coach can work together to learn which strategies work best for you and to try to make strategies that are more challenging easier to use.


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022





A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

ESDM-informed caregiver coaching is a therapy developed from an evidence-based form of behavioral therapy called ESDM that uses principles of Applied Behavior Analysis (ABA) to promote language, social interaction, and behavioral regulation. During each coaching session, the therapist will:

- Check in with you to see how things are going with your child.
- Briefly talk about the strategies to be learned and practiced during that coaching session.
- Give you feedback as you work with your child trying the strategy and other techniques.
- Towards the end of the appointment, you and the therapist will talk about specific things to try during the next week.

#### **Assessment Visits and Questionnaires**

You and your child will complete several questionnaires and activities remotely to help us understand how your child is progressing in paying attention to things going on around them, their social and language skills, and their behavior. It is important that you, not some other caretaker, complete the questionnaires and attend the remote visits so that we can see and measure the changes in your child over time as accurately as possible.

Remote assessment visits will be held via Zoom and will take around 1-2 hours. The activities are described below. They will be repeated 1 week after completing 8 weeks of ESDM-informed caregiver coaching.

#### Questionnaires and Interviews

- You will be asked to complete a set of questionnaires (sent electronically), which include questions about your child's social skills, language, emotional expression, interests, and other behaviors, such as sleep habits. Some of these will also ask how you and your child are feeling and doing, and about your experiences in the study.
- There will also be parent interviews where we will ask you about the behaviors that you observe your child doing regularly in your home where we can't observe your child ourselves.

#### Assessment of social interaction, communication, and attention

Your child will participate in activities that involve playing with toys and observing how he/she responds to you. Some of these activities will be recorded through the Duke Zoom platform. The recordings are used for data collection, data monitoring and review of parent-child interactions and the clinician's prompts. For privacy and data integrity reasons, session recordings cannot be shared with participants and must remain stored with the study records.

| Parent | /Guardian | Initials |
|--------|-----------|----------|





A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

- In the event that recording Zoom sessions is not possible due to connectivity issues, the study team will provide you with instructions for how to record coaching and parent-child interaction sessions using your own device. The study team will create a unique link for you to upload the videos a secure, encrypted, Duke Health affiliated server (Duke Box) that only the study team has access to.
- Other assessments of social interaction and communication. We will record these interactions so we can go back and count how often specific behaviors occur to get more precise measurements that might show change over time
  - We will observe and videotape how your child naturally plays with you and a specific set of toys at home.
  - You and your child may view a set of short engaging videos on an iPhone or iPad, and the camera will record your child's facial expressions and responses to the videos. You may use your own iPhone/iPad, or a borrowed one.

**At 16 weeks**, we will ask you to complete follow-up assessments, including an interview about your child's behavior and electronic questionnaires.

If your child is reporting symptoms that may require medical attention, the study doctor may recommend that your child receive certain procedures or tests through your child's doctor, even though the tests are not listed as part of the study. You can refuse the study doctor's recommendations for these things, but refusal may affect you and your child's participation in the study and could result in you and your child being taken out of the study.

#### **Future Contact**

If you enroll your child in the Duke ACE program you may receive the following information occasionally:

- Email requests to inform us of any changes in your contact information (address, e-mail address, and/or phone number),
- Newsletters to update you on ongoing activities of the Duke ACE Center,


- Holiday and birthday cards,
- Invitations to special community events hosted by the Center (such as virtual music events, sports clinics, and artwork contests),
- Information about other research-related opportunities, including the Registry for Autism Research.

#### **Contact with the A+ Treatment Study Team**

The study will use email (acetreatment@duke.edu) to communicate with you about visit scheduling and follow-ups as needed. Because using your personal e-mail does not provide a

| Parent/Guardian | Initials |
|-----------------|----------|



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

completely secure and confidential means of communication, please do not use it if you wish to keep your communication private. Instead, let us know and we will communicate with you through Duke secure mail and telephone. You may also call the study coordinator or other staff covering for the coordinator at (919)-681-0017, which is a secure phone line.

# Video and Audio and Sensor Recording of Assessments

Audio and video recordings of assessments of you and your child (e.g., in behavioral, play-based activities, or interviews conducted with you and/or your child) and sensor information from the iPad or iPhone collected while your child is watching the movies, such as audio and video recordings, including calling your child's name) will be collected, stored, and used for data analysis and for quality monitoring of the assessments. If you agree, these recordings may also be used for training or educational purposes. Please indicate your choices below.

Yes: I give permission for images/videos of myself and/or my child to be used

for educational and training purposes.

**No:** I DO NOT give permission for images/videos of myself and/or my child to be

used for educational and training purposes.

Yes: I give permission to have images/videos of myself and/or my child to be

used in scientific meetings, articles, and research publications.

**No:** I DO NOTgive permission to have images/videos of myself and/or my child to be

used in scientific meetings, articles, and research publications.

**Privacy at home:** This study involves taking video and audio recordings while you are participating in coaching and parent-child interactions. For the study visits and any study-related phone calls/interviews, we ask that you identify places where you can comfortably speak to our team, and where you can engage in study activities without disruptions, as these could be captured on camera/recordings.

#### **HOW LONG WILL I BE IN THIS STUDY?**

Participation in the study is expected to require 10 weeks plus a follow-up assessment at 16 weeks.

#### WHAT ARE THE RISKS OF THE STUDY?

There is a possibility that you or your child may become frustrated during study tasks. We will try to make the tasks and task directions as easy as possible. Your child can take as many

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

breaks as he/she needs during assessments. Some of the questions we will ask you or your child as part of this study may make you or your child feel uncomfortable. You or your child may refuse to answer any of the questions and you or your child may take a break at any time during the study. You or your child may stop your participation in this study at any time.

There is also the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

## Risks related to your child's ASD and ADHD

Your child may experience a worsening of symptoms that may be because of their condition alone, or because of a lot of other factors that may not be related to this study. In cases of severe worsening of symptoms that place your child or those around him/her at risk, your child may require inpatient hospitalization. If the study doctor feels that your child is at serious risk for hurting him/herself or others, he/she can ask a judge to allow your child to be hospitalized against your and/or your child's will.

If your child is on any medication, please speak with your child's doctor about the risks of those medications.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you and your child agree to take part in this study, your child may benefit by receiving some of the diagnostic and cognitive evaluations that are conducted as part of this study. Your family could also benefit from the ESDM-informed caregiver coaching and learning how to use strategies for promoting social skills, language, and behavioral regulation.

There are potential benefits for receiving a caregiver-coaching behavioral therapy along with other behavioral assessments as previously mentioned. Finally, we also hope that in the future the information learned from this study will benefit other people with both ASD and ADHD.

#### WHAT ALTERNATIVES ARE THERE TO PARTICIPATION IN THIS STUDY?

Instead of being in this study, you and your child have the following alternatives:


- Other early intervention therapy for ASD
- Other behavior therapy for ADHD in young children
- Have your child try medicine for associated symptoms, such as anxiety or irritability

Please talk to your child's doctor about these and perhaps other options.



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

#### WILL MY CHILD'S INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. This study will collect information that might directly identify you and your child, such as names, dates of birth, addresses and health related information. We understand that information about you and your child's health is personal, and we are committed to protecting the privacy of that information. We will do our best to make sure that information about you and your child is kept confidential, but we cannot guarantee total confidentiality. You and your child's personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. Collaborators include individuals who are not part of Duke University. We will share only the minimum information in order to conduct the research. You and your child's personal information may also be given out if required by U.S. or State law. Examples of information that we are legally required to disclose include abuse or neglect of a child.

As part of the study, results of your child's study-related data and procedures may be reported to the NIH and its affiliates. In addition, your child's records may be reviewed in order to meet federal or state regulations. Reviewers may include representatives from the Food and Drug Administration (FDA), representatives and affiliates of the NIH, and the Duke University Health System Institutional Review board, and others as appropriate. If any of these groups review your child's research record, they may need to review your child's entire medical records.

The Duke ACE Center will use a third-party web-based application from NCS Pearson, Inc. (Q-Global) to administer and score the responses for some assessments in this research program. To properly score this assessments, information including your child's gender, date of birth, and his/her study ID will be entered along with assessment responses. Remote questionnaire completion also requires a parent/guardian's name and email address to be entered in to Q-Global. The minimal amount of information will be submitted to Q-Global for purposes of administering and accurately scoring the assessments. The information provided to Q-Global is subject to their terms of use. Data is encrypted using industry-standard SSL technology and compliant with established HIPAA Security Regulations as well as changes to HITECH Act effective March 2013 which applies to Business Associates to health care providers. NCS Pearson, Inc. shall not use or disclose PHI other than permitted or required by the HIPAA Rules or as required by law. NCS Pearson, Inc. may use data in de-identified form during the testing process for internal quality control, operations management, security, and research to enhance, develop and improve tests and testing processes.

De-identified data means that data cannot be identified as belonging to any individual and specifically meets the de-identification standard as required by HIPAA. As with any website platform or software, there may be potential security risks and Duke cannot guarantee that the


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

website is free of risk. If the data are further disclosed by Q-Global, they are no longer covered by the Duke privacy protections.

Except when required by law, and as otherwise explained in this consent document, you or your child will not be identified by name, address, telephone number, or any other direct personal identifier in records disclosed outside of Duke University Health System (DUHS). All data can only be accessed by a secure password which will be locked away by authorized personnel. The database will be stored on a secure server at the Duke School of Medicine. Study team members are required to log in with a unique username and password to access the study database. Before being granted access to the study database, staff complete training on protecting confidentiality and sign confidentiality agreements. The database will include all the information that we collect during the course of the study and it will also include information such as your child's date of birth, gender, and date of each study visit. It also will contain your child's name and contact information in a dashboard. All hard copies of your child's records will be kept in locked file cabinets. Only people who need access to your child's data to do their job will have access to it. Any paper records will be stored in locked office.

This project is part of a larger set of projects that are part of the Duke Autism Center of Excellence funded by the National Institute of Child Health and Human Development. The data that we collect for this study will be shared with other researchers at Duke, including researchers working with Duke Center for Autism investigators. Combining data across many research projects and other studies allows us to learn more about early childhood development. Your data may also be shared with qualified researchers outside of Duke for the purpose of research only.

Some research information such as psychological assessment reports will be available to you upon your request.

The study results will be retained in your child's research record for six years after the study is completed or until your child reaches the age of 21, whichever is longer. At that time either the research information not already in your child's medical record will be destroyed or information identifying your child will be removed from such study results at DUHS. Any research information in your child's medical record will be kept indefinitely.

This information may be further disclosed by NIMH (National Institute of Mental Health), the funding agency of this study. If disclosed by the funding agency, the information is no longer covered by federal privacy regulations. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations. NIMH is a part of the NIH.

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 09/20/2021 IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your and your child's name or other personal information will not be revealed, unless you have given us permission to do this through another separate permission form.

Some people or groups who receive your and your child's health information might not have to follow the same privacy rules. Once your and your child's information is shared outside of Duke, we cannot guarantee that it will remain private. If you decide to share your or your child's private information with anyone not involved in the study, the federal law designed to protect your and your child's health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

#### **NDAR**

Data from this study may be submitted to the National Data for Autism Research (NDAR). NDAR is a data repository run by the NIMH that allows researchers studying children's health to collect and share de-identified information with each other. A data repository is a large database where information from many studies is stored and managed. De-identified information means that all personal information (such as name, address, and phone number) is removed and replaced with a code number. With an easier way to share, researchers hope to learn new and important things about children's health more quickly than before.

During and after the study, we will send de-identified information to NDAR. Other researchers nationwide can then file an application with the NIMH to obtain access to your or your child's de-identified study data for research purposes. Experts at the NIMH who know how to protect health and science information will look at every request carefully to minimize risks to your privacy.

You may not benefit directly from allowing your information to be shared with NDAR. The information provided to NDAR may help researchers around the world treat future children and adults with mental illnesses so that they have better outcomes. NIMH will also report to Congress and on its web site about the different studies that researchers are conducting using NDAR data. However, you will not be contacted directly about the data you contributed to NDAR.

You may decide now or later that you do not want to share your or your child's information using NDAR. If so, contact Dr. Dawson and she or a research study staff member will tell NDAR, which can stop sharing the research information. However, NDAR cannot take back information that was shared before you changed your mind. If you would like more information about NDAR, this is available on-line at <a href="http://data-archive.nimh.gov">http://data-archive.nimh.gov</a>.

| | Parent/Guardian | Initials |
|---------------|------------------|----------|
| . ago . o o | . aroni oaaralan | |



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

If you agree or have agreed to store your data in the **Duke Center for Autism Data Sharing Repository (DSR)**, we will use your data from previous Duke Center for Autism studies as part of this research study to help prevent you from doing duplicate assessments. If you sign or have signed a DSR consent form, we will also add the data from this study to the DSR database for future use. If you have questions about the DSR or would like a copy of the consent form, please ask the staff member reviewing this consent form with you or contact autismresearch@duke.edu.

# **Certificate of Confidentiality**

The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your privacy. With this Certificate, the investigators may not disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use. Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:

- 1) There is a law that requires disclosure (such as to report child abuse or communicable diseases but not for legal proceedings);
- 2) You have consented to the disclosure, including for your medical treatment; or
- 3) The research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project or for information that is required by the FDA.

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy.

Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.


DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

# WHAT ARE THE COSTS TO YOU?

There will be no additional costs to you or your child as a result of being in this study. However, routine medical care received at Duke for your child's condition (care your child would have received whether or not your child was in this study) will be charged to you or your insurance company. You may wish to contact your insurance company to discuss this further.

#### WHAT ABOUT COMPENSATION?

You and your child will be compensated up to a total of \$550 for participating in this study. You will be reimbursed \$50 for your participation in the assessments and coaching at each study time point (Baseline, and weekly through Week 9). Participants will be compensated (\$50) for completing assessments at week 16.

Payment received as compensation for participation in research is considered taxable income to the research subject. If payment to an individual totals \$600 or more in any one calendar year, Duke University is required to report this information to the Internal Revenue Service (IRS). Research subject payments to a non-employee of Duke University adding up to \$600 or more during any calendar year will result in a 1099 (Miscellaneous Income) form being issued to the individual and a copy sent to the IRS.

#### WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that your child is injured as a result of your child's participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your Duke physicians to provide monetary compensation or free medical care to you in the event of a study-related injury.

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, contact Dr. Franz at (919) 681-0023 or (919)-627-1652 for Dr. Chandrasekhar (another doctor on the study) after hours and on weekends and holidays.

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You and your child may choose not to be in the study, or, if you and your child agree to be in the study, you or your child may withdraw from the study at any time. If you or your child withdraw from the study, no new data about your child will be collected for study purposes other than data needed to keep track of your child's withdrawal, unless the data concern an adverse event related to the study. All data that have already been collected for study purposes, and any new information about an adverse event related to the study, will be

DUHS |RB IRB NUMBER: Pro00085179 IRB REFERENCE DATE: 09/20/2021 IRB EXPIRATION DATE: 04/04/2022

 Parent/Guardian Initials\_\_\_\_\_



A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

included in the research database. All data that have already been collected will be kept solely for study purposes and will be sent to the study sponsor.

You or your child's decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you and your child are entitled, and will not affect your child's access to health care at Duke. Signing this consent form is not a condition for receiving any medical care outside the study. However, if you or your child decides to stop participating in the study, we encourage you to talk to your child's doctor first. If you do decide to withdraw, we ask that you contact Dr. Franz in writing and let her know that you are withdrawing from the study. Her email address is: <a href="mailto:lauren.franz@duke.edu">lauren.franz@duke.edu</a>, and her phone number is: (919) 681-0023.

If you use email please be aware that you may be at potential risk for a loss of confidentiality because email is not a secure means of communication.

If for any reason you decide to discontinue the behavioral coaching, but are willing to complete the other measures of the study, the study doctor may ask you and your child to complete the tests that would ordinarily occur when a person completes the study.

Your child's study doctor may decide to discontinue your child's participation in this study if your child's condition gets worse, or if your child's study doctor determines that it is no longer in your child's best interest to continue. The funding agency or regulatory agencies may stop this study at any time without your or your child's consent. Reasons why this might occur include because your child has failed to follow instructions, or because the entire study has been stopped. If this occurs, you will be notified and your child's study doctor will discuss other options with you.

If you do not sign this consent form and your child is a Duke patient, your child will continue to receive care from your healthcare provider, but not as a part of this study.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify your child. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, contact Dr. Franz at (919) 681-0023 or (919)-627-1652 for Dr. Chandrasekhar after hours and on weekends and holidays.

DUHS RB
IRB NUMBER: Pro00085179
IRB REFERENCE DATE: 09/20/2021
IRB EXPIRATION DATE: 04/04/2022

Form M0345



# Consent to Participate in a Research Study

A+ Treatment/Feasibility (Sub-study): Feasibility trial of adapted ESDM-informed caregiver coaching delivered remotely for children with ASD and ADHD

**Duke Autism Center of Excellence Research Program** 

For questions about your or your child's rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.

#### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask the questions I have, and my questions have been answered to my satisfaction. I have been told whom to contact if I have additional questions. I have read this consent form and agree to participate and allow my child to be in this study with the understanding that I may withdraw him/her or myself at any time. We have discussed the study with my child, who agrees to be in the study. I have been told that I will receive a copy of this consent form, which will be sent to the email address (es) I choose to include below."

| Signature of Parent/Guardian #1 | Date | Time |
|-------------------------------------------------|------|------|
| Name of Parent/Guardian #1 | | |
| Signature of Parent/Guardian #2 (if applicable) | Date | Time |
| Name of Parent/Guardian #2 (if applicable) | | |
| Signature of Person Obtaining Consent | Date | Time |
| Name of Person Obtaining Consent | | |
| email address #1:email address#2(optional): | | |